CLINICAL TRIAL: NCT03571854
Title: Comparison of Pressure-controlled Ventilation-volume Guaranteed Mode With Volume Controlled Ventilation in Prone Position During Lumbar Spine Surgery.
Brief Title: The Effect of Pressure-controlled Ventilation-volume Guaranteed Mode
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-I036
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PCV-VG (Experimental): Pressure controlled ventilation-volume guaranteed
  Interventions: Device: Group PCV-VG
- Group VCV (Active Comparator): Volume controlled ventilation
  Interventions: Device: Group VCV

INTERVENTIONS:
Device: Group PCV-VG — Pressure controlled ventilation-volume guaranteed
  Arms: Group PCV-VG
Device: Group VCV — Volume controlled ventilation
  Arms: Group VCV

SUMMARY:
The anesthetized patient is turned to the prone position during lumbar spine surgery. The dynamic compliance of lung usually decreases and peak airway pressure increases during the surgery.

A new ventilation mode, pressure-controlled ventilation with volume guaranteed mode (PCV-VG) has been recently introduced. The ventilator compares the tidal volume of the previous breath and automatically regulates the pressure up or down to achieve the set tidal volume.

This prospective, randomized study is designed to compare the effect of PCV-VG and volume-controlled ventilation (VCV) on peak airway pressure, lung compliance and hemodynamic variables.

DETAILED DESCRIPTION:
1. Total 34 patients with American Society of Anesthesiologists physical status I-III who underwent lumbar spine surgery in prone position were enrolled.
2. All patients fasted for 8 hours before the surgery and were premedicated with intramuscular glycopyrrolate 0.2 mg. Anesthesia was induced with remifentanil (0.1-0.2 ug/kg/min), propofol (1.5-2 mg/kg) and rocuronium (0.6 mg.kg) and maintained with sevoflurane (2.0-2.5 vol%) in inspired oxygen fraction with 0.5, remifentanil (0.05-0.3 ug/kg/min) and vecuronium (0.03-0.05 mg/kg/hr).
3. A 20 G catheter was inserted into the radial artery to monitor continuous arterial pressure and hemodynamic variables (cardiac output, cardiac index, stroke volume, stroke volume index, and stroke volume variation) monitoring.
4. All patients were ventilated with a Datex-Ohmeda Ventilator (S/5 AVANCE). Patients were randomized to receive either PCV-VG (n=17) or VCV (n=17) mode. The tidal volume in both group were set to deliver 8 mL/kg of ideal body weight. The respiratory rate (RR) was adjust to maintain end tidal CO2 (ETCO2) 33-38 mmHg.
5. Hemodynamic variables (mean blood pressure, heart rate, cardiac output, cardiac index, stroke volume, stroke volume index, and stroke volume variation) , respiratory variables (saturation, RR, ETCO2, peak airway pressure, mean airway pressure and lung dynamic compliance) and arterial gas analyses were recorded at 4 stages: (1) 15 minutes after induction in supine position, (2) 30 minutes after turning the patient to the prone position, (3) 60 minutes after turning the patient to the prone position, (4) 15 minutes after turning the patient to supine position at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for lumbar spine surgery with the prone position
* American Society of Anesthesiologists physical status I-III

Exclusion Criteria:

* Age under 20 years old or over 70 years old
* Body mass index > 30 kg/m2
* Systolic blood pressure < 100 mmHg
* Heart rate < 60 bpm
* Uncompensated cardiac disease
* FEV1 < 60%
* Hypoxemia (PaO2 < 60 mmHg or oxygen saturation < 90%)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-07-21 (Estimated); Study Completion 2018-07-28 (Estimated)

PRIMARY OUTCOMES:
Peak airway pressure | About 2-3 hours through the surgery
  The highest level of pressure applied to the lungs during inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Eun Young Park, MD, Study Director — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Dongan-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jo YY, Kim JY, Kwak YL, Kim YB, Kwak HJ. The effect of pressure-controlled ventilation on pulmonary mechanics in the prone position during posterior lumbar spine surgery: a comparison with volume-controlled ventilation. J Neurosurg Anesthesiol. 2012 Jan;24(1):14-8. doi: 10.1097/ANA.0b013e31822c6523. PMID 21897297
- [Background] Pu J, Liu Z, Yang L, Wang Y, Jiang J. Applications of pressure control ventilation volume guaranteed during one-lung ventilation in thoracic surgery. Int J Clin Exp Med. 2014 Apr 15;7(4):1094-8. eCollection 2014. PMID 24955188
- [Background] Dion JM, McKee C, Tobias JD, Sohner P, Herz D, Teich S, Rice J, Barry ND, Michalsky M. Ventilation during laparoscopic-assisted bariatric surgery: volume-controlled, pressure-controlled or volume-guaranteed pressure-regulated modes. Int J Clin Exp Med. 2014 Aug 15;7(8):2242-7. eCollection 2014. PMID 25232415
- [Background] Keszler M. Volume-targeted ventilation. Early Hum Dev. 2006 Dec;82(12):811-8. doi: 10.1016/j.earlhumdev.2006.09.008. Epub 2006 Oct 27. PMID 17069993
- [Background] Song SY, Jung JY, Cho MS, Kim JH, Ryu TH, Kim BI. Volume-controlled versus pressure-controlled ventilation-volume guaranteed mode during one-lung ventilation. Korean J Anesthesiol. 2014 Oct;67(4):258-63. doi: 10.4097/kjae.2014.67.4.258. Epub 2014 Oct 27. PMID 25368784
- [Derived] Lee JM, Lee SK, Kim KM, Kim YJ, Park EY. Comparison of volume-controlled ventilation mode and pressure-controlled ventilation with volume-guaranteed mode in the prone position during lumbar spine surgery. BMC Anesthesiol. 2019 Jul 27;19(1):133. doi: 10.1186/s12871-019-0806-7. PMID 31351445